CLINICAL TRIAL: NCT06933160
Title: Promotion of Exercise for Multiple Sclerosis Through Physical Therapy (PromPT)
Brief Title: Promotion of Exercise Through Physical Therapy for Multiple Sclerosis: A Pilot Study
Acronym: PromPT-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Dominique Kinnett-Hopkins, Assistant Professor of Kinesiology, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00266361; 1R03HD111005-01A1 (NIH)
Record Dates: First submitted 2025-04-05; First posted 2025-04-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; physical activity; exercise; physical therapy
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): The experimental intervention is a 24-week progressive exercise intervention in which participants are supported through six physical therapy visits and are provided with educational material based on social cognitive theory. The individual sessions will provide tailored support for increasing physical activity behavior towards the recommended guidelines of 2-3 moderate aerobic activity sessions and two strength-training sessions per week. There are no drugs involved in the intervention.
  Interventions: Behavioral: PromPT-MS
- Waitlist Control (No Intervention): 24-week waitlist control condition

INTERVENTIONS:
Behavioral: PromPT-MS — The experimental intervention is a 24-week progressive exercise intervention in which participants are supported through six physical therapy visits and are provided with educational material based on social cognitive theory. The individual sessions will provide tailored support for increasing physical activity behavior towards the recommended guidelines of 2-3 moderate aerobic activity sessions and two strength-training sessions per week. There are no drugs involved in the intervention.
  Arms: Experimental

SUMMARY:
Physical activity and exercise help manage symptoms like fatigue in people living with multiple sclerosis (MS). Despite research supporting physical activity participation, people with MS are often insufficiently active to reach health benefits. Promotional efforts that are sustainable within the United States healthcare system are needed. This project is a pilot randomized controlled trial examining the feasibility of a consultative physical therapy intervention for increasing physical activity engagement.

DETAILED DESCRIPTION:
Multiple sclerosis is a debilitating disease usually diagnosed between the ages of 20 and 49 years with no curative options, resulting in a focus on rehabilitation strategies to manage symptoms, restore function, and improve quality of life. Physical activity, particularly exercise training, is considered one of the best rehabilitation strategies for comprehensive multiple sclerosis management. Despite strong evidence of the safety and benefits of physical activity and exercise in this population, persons with multiple sclerosis do not engage in sufficient levels of physical activity. Physical therapists are well positioned and have the expertise to facilitate physical activity and exercise participation for persons with multiple sclerosis. However, physical therapy is underutilized, particularly in people with more mild multiple sclerosis symptoms, when the best results may be achieved. A proactive physical therapy delivery model may help persons with multiple sclerosis increase and maintain their physical activity and exercise behaviors. The proposed study involves 1) a randomized controlled trial to evaluate outcomes of feasibility in the four metrics of process, resources, management, and scientific outcomes, and 2) an assessment of the immediate and sustained treatment effect of the physical therapy model compared to a waitlist control on accelerometer-measured physical activity. The feasibility trial will be conducted with a sample of 40 persons with multiple sclerosis randomized to either the intervention or waitlist control group. Participants will complete assessments at baseline, post-intervention (6 months), and follow-up (10 months). Participants will complete a formative evaluation, including surveys and one-on-one semi-structured interviews, to assess satisfaction, acceptability, feasibility, and appropriateness of the physical therapy delivery model. The proposed feasibility study, interviews, and implementation assessments will directly lead to the submission of an R01 to test the efficacy of an appropriately powered randomized controlled trial and to identify context-specific barriers and facilitators to the successful uptake of this physical therapy model in clinical settings. The dissemination of the results of this feasibility study can lead to improvements in physical therapy delivery for persons with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS
* 18 years and older
* Able to read and speak English sufficiently to allow for informed consent and active participation in the intervention sessions
* Relapse free for the past 30 days
* Willingness to attend all study visits and PT sessions for the duration of study
* Access to a smartphone
* Not sufficiently active as measured by the Godin Leisure Time Exercise Questionnaire score <24
* Patient Determined Disease Steps score 0-3 or the ability to ambulate either independently or with the use of a cane (or similar device) for at least 75% of the time at baseline
* Less than 2 affirmative on the physical activity readiness questionnaire

Exclusion Criteria:

* Inability to provide informed consent (e.g., cognitive impairment, unable to sufficiently communicate in English)
* Unable to attend study visits
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-measured moderate-to-vigorous physical activity | From enrolment to end of treatment at 24 weeks
  The duration (in minutes per day) of moderate-to-vigorous physical activity (MVPA) will be assessed using a waist-worn accelerometer (ActiGraph model GT3X+). Participants will wear the accelerometer attached to a belt around their waist during waking hours over a 7-day period. A greater duration of MVPA indicates a higher level of physical activity.

SECONDARY OUTCOMES:
Total physical activity | From enrolment to end of treatment at 24 weeks
  The duration (in minutes per day) of physical activity (light, moderate, and vigorous activity) will be assessed using a waist-worn accelerometer (ActiGraph model GT3X+). Participants will wear the accelerometer attached to a belt around their waist during waking hours over a 7-day period. A greater duration of physical activity indicates a higher level of physical activity.
Fatigue | From enrolment to end of treatment at 24 weeks
  PROMIS Fatigue CAT
Physical Function | From enrolment to end of treatment at 24 weeks
  PROMIS Physical Function CAT
Exercise Self-efficacy | From enrolment to end of treatment at 24 weeks
  Exercise Self-efficacy scale

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Kinnett-Hopkins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No